CLINICAL TRIAL: NCT05882032
Title: A Phase 1, Multicenter, Parallel, Single-Dose, Open-Label, Single-Period Study of LY3502970 in Participants With Normal Hepatic Function and Participants With Mild, Moderate, or Severe Hepatic Impairment
Brief Title: A Study of LY3502970 in Participants With Impaired and Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18624; J2A-MC-GZPB (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Hepatic Insufficiency
Keywords: LY3502970; Pharmacokinetics Hepatic Impairment; GLP-1 Receptor Non-peptide agonist (GLP-1 NPA)
MeSH Terms: conditions — Hepatic Insufficiency | interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3502970 (Mild Hepatic Impairment) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970
- LY3502970 (Moderate Hepatic Impairment) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970
- LY3502970 (Severe Hepatic Impairment) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970
- LY3502970 (Normal Hepatic Function) (Experimental): LY3502970 administered orally.
  Interventions: Drug: LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered orally.

SUMMARY:
The main purpose of this study is to measure how much of LY3502970 gets into the bloodstream and how long it takes the body to eliminate it in participants with mild, moderate and severe impaired liver function compared to participants with normal liver function. The safety and tolerability of LY3502970 will also be evaluated. The study may last up to 6 weeks for each participant including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with body weight of at least 45 kilograms and a body mass index of 18.5 to 40.0 kilograms per meter squared (kg/m²).
* Both healthy individuals and individuals with hepatic impairment classified as Child-Pugh Score A, B, C that is mild, moderate, or severe impairment, respectively, liver disease can participate who are considered acceptable for participation in this study by the investigator.
* Participants must have a diagnosis of chronic hepatic impairment for more than 6 months per physician diagnosis and standard of care practice, with no clinically significant changes within 15 days prior to study intervention administration.
* Participants may have mild stable baseline medical conditions for which neither the condition nor treatments received would negatively impact the health of the participant or study conduct.
* Have acceptable BP and pulse rate, as determined by the investigator at screening.
* No significant history of spontaneous or ethanol induced hypoglycemia.
* Participants with Mild to Severe Hepatic Impairment who have a hemoglobin level of at least 8.5 grams/deciliter.
* Participants with both T2DM and Hepatic Impairment have T2DM controlled with diet or exercise alone or on stable doses of anti-diabetic medications metformin or sulfonylureas, for at least 8 weeks prior to screening.
* Participants with both T2DM and Hepatic Impairment have a hemoglobin A1c greater than or equal to 5.0% and less than or equal to 11.0% at the screening visit.
* Participants with both T2DM and Hepatic Impairment have clinical laboratory test results within normal range or deemed clinically insignificant by the investigator. Abnormalities of serum glucose, serum lipids, urinary glucose, and urinary protein consistent with T2DM are acceptable.

Exclusion Criteria:

* Have significant history of, or current, cardiovascular, respiratory, hepatic (applies to Group 1 only), renal, GI, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs.
* Have a history or presence of pancreatitis, elevation in serum amylase or lipase (greater than 1.5-fold ULN) or GI disorder or any GI disease, which impacts gastric emptying.
* Have any abnormality in the 12-lead ECG at screening.
* Have severe atopy or have a history of clinically significant multiple or severe drug allergies or severe post treatment hypersensitivity reactions.
* Have a history of, or current psychiatric disorders.
* Women who are pregnant, intend to become pregnant or are breastfeeding a child are not eligible to participate.
* Have taken any glucose-lowering medications other than metformin, sulfonylureas, and insulin, in the past 6 weeks or 5 half-lives (whichever is longer) prior to planned dosing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the concentration versus time curve from time zero to infinity (AUC0-∞) of LY3502970 | Predose up to 96 hours postdose
  PK: AUC0-∞ of LY3502970
PK: Area under the concentration versus time curve from time zero to last time point (AUC0-tlast) of LY3502970 | Predose up to 96 hours postdose
  PK: AUC0-tlast of LY3502970
PK: Maximum observed concentration (Cmax) of LY3502970 | Predose up to 96 hours postdose
  PK: Cmax of LY3502970

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3502970 in Participants With Impaired and Normal Liver Function — https://trials.lilly.com/en-US/trial/407541